CLINICAL TRIAL: NCT05119933
Title: A Phase 1/2, Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of YL-15293 in Subjects With Advanced Solid Tumors With a KRAS G12C Mutation
Brief Title: A Phase 1/2, Study of YL-15293 in Subjects With Advanced Solid Tumors With a KRAS G12C Mutation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Collaborators: Yingli Pharma US, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-15293-001
Record Dates: First submitted 2021-11-11; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-09

CONDITIONS: Advanced Solid Tumor
Keywords: with a KRAS G12C mutation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YL-15293 (Experimental): After a screening period of approximately 28 days, eligible patients will receive oral YL-15293 once daily until documented disease progression, unacceptable AEs, intercurrent illness prevents further administrations of study treatment, investigator's decision to withdraw the patient, the patient withdraws consent, pregnancy of the patient, or for administrative reasons. Following the end of treatment, patients will continue to be followed for safety for 30 days. Patients who permanently discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.
  Interventions: Drug: YL-15293

INTERVENTIONS:
Drug: YL-15293 — After a screening period of approximately 28 days, eligible patients will receive oral YL-15293 once daily until documented disease progression, unacceptable AEs, intercurrent illness prevents further administrations of study treatment, investigator's decision to withdraw the patient, the patient withdraws consent, pregnancy of the patient, or for administrative reasons (see Section 7.1). Following the end of treatment, patients will continue to be followed for safety for 30 days. Patients who permanently discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.

SUMMARY:
This is a Phase 1/2, open-label, multicenter study designed to evaluate the maximum tolerated, safety, tolerability and PK of oral YY-15293 in patients with advanced solid tumors with a KRAS G12C mutation, to confirm the recommended phase 2 dose of YY-15293, and to obtain preliminary efficacy information in patients with advanced non-small cell lung cancer (NSCLC) with a KRAS G12C mutation.

DETAILED DESCRIPTION:
The study will be conducted in the United States of America (USA) and China to provide safety, efficacy and PK data from these regions. A dose escalation part 1 will be conducted to determine the MTD, DLT's, and part 2 will confirm the safety/tolerability of the recommended Phase 2 dose (RP2D), of YL-15293 given once daily, in patients with advanced NSCLC to obtain preliminary efficacy information. PK samplings at Cycle 1, Day 1 and at steady-state conditions (Cycle 1, Day 28) will be performed. PD evaluations will occur at cycle 1 and cycle 2.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for participation in this trial, the patient must meet all the following criteria:

  1. Part 1 only - metastatic or locally advanced solid tumor malignancies positive for KRAS G12C that has progressed on, is refractory to, intolerant to, or for which there is no curative standard of care therapy.

     Part 2 only - metastatic or locally advanced KRAS G12C NSCLC for patients for whom there is no curative standard of care therapy.
  2. Measurable disease with at least 1 lesion amenable to response assessment per RECIST 1.1.
  3. Demonstrate adequate organ function as defined below. All screening laboratories should be performed within 14 days of treatment initiation.
  4. Has a performance status of 0-2 on the ECOG Performance scale.
  5. Life expectancy more than12 weeks at baseline.
  6. Women of childbearing potential must have negative serum or urine pregnancy test within 72 hours prior to receiving the first study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  7. For women of childbearing potential, must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and 120 days following last day study drug administration.
  8. Male patients of childbearing potential must be surgically sterile, or must agree to use adequate method of contraception during the study and at least 120 days following the last day of study drug administration.
  9. Age more than18 years at screening.
  10. Able and willing to provide written informed consent and to follow study instructions.

Exclusion Criteria:

* Patients are excluded from the study if any of the following criteria apply:

The patient will be excluded from participating in the trial if meet any of the following:

1. Patient has disease that is suitable for therapy administered with curative intent.
2. Subjects who have received prior treatment with KRAS G12C targeted agents.
3. Subjects who have received 4 or more lines of prior therapy.

The patient will be excluded from participating in the trial if meet any of the following:

1. Patient has disease that is suitable for therapy administered with curative intent.
2. Subjects who have received prior treatment with KRAS G12C targeted agents or pan-KRAS inhibitors.
3. Subjects who have received 4 or more lines of prior therapy.
4. Central nervous system (CNS) involvement with tumor.
5. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment.
6. Unresolved toxicities from prior therapy, defined as having not resolved to NCI CTCAE v.5.0 Grade 0 or 1, with exception of endocrinopathies from prior therapy and successfully treated (such as hypothyroidism), as well as alopecia and vitiligo.
7. Patient has an active infection requiring systemic therapy.
8. Patients who have known active HIV, Hepatitis or Hepatitis or active COVID-19 infection. (Patients who have been vaccinated against Hepatitis B and who are positive only for the Hepatitis B surface antibody are permitted to participate in the study). Subjects who are positive for HIV or hepatitis B or C virus must be tested for and have an undetectable viral load.
9. Patients with unstable/inadequate cardiac function:

   New York Heart Association Class 3 or 4 congestive heart failure, Uncontrolled hypertension, Acute coronary syndrome within 6 months, Clinically significant cardiac arrhythmia, Mean QTC interval corrected for heart rate >500ms.
10. Patient has a history of interstitial lung disease.
11. Current active additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
12. Participation in another clinical trial of an investigational agent within 30 days of screening.
13. Patient has known psychiatric, substance abuse or other disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the investigator.
14. Patients who are pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-11-09 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) | Throughout the study for approximately 2 years
  The overall response rate (ORR) will be estimated based on the proportion of evaluable patients whose overall response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1.

SECONDARY OUTCOMES:
Progression free survival, PFS | Throughout the study for approximately 2 years
  PFS, defined as the time from the first dose of study treatment to first
Overall survival, OS | Throughout the study for approximately 2 years
  The time from randomization to death for any reason
Disease control rate, DCR | Throughout the study for approximately 2 years
  The percentage of cases with remission (PR+CR) and stable lesions (SD) after treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Innovative Clinical Research Institute, Whittier, California
  - The Tisch Cancer Institute Mount Sinai Health System Icahn School of Medicine at Mount Sinai, New York, New York
  - Oncology Consultants, Houston, Texas